CLINICAL TRIAL: NCT05075733
Title: The Current Scope of Practice of Today's Hepatopancreatobiliary Surgeons: A Survey of Americas Hepato-Pancreato-Biliary Association Members
Brief Title: Current Scope of Practice of Today's Hepatopancreatobiliary Surgeons: A Survey of AHPBA Members
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: IRBNET#0000000
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Scope of Practice of Today's Hepatopancreatobiliary Surgeons
Keywords: survey; AHPBA
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey was sent to all the Americas Hepato-Pancreato-Biliary Association's members

SUMMARY:
The development of multiple training pathways to foster competent hepatopancreatobiliary (HPB) surgeons has led to a diverse group of surgical subspecialists. The objective of our study was to determine the current scope of practice of today's HPB surgeons. An online survey was sent to all the Americas Hepato-Pancreato-Biliary Association's members to assess the current scope of practice of today's HPB surgeons. We found very few surgeons run a solo HPB practice, so changes may be needed in HPB training to provide uniformity and enhance the scope of practice for future HPB surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Member of Americas Hepato-Pancreato-Biliary Association

Exclusion Criteria:

* No or non-functioning email address

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Member of Americas Hepato-Pancreato-Biliary Association
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Survey outcome 1 | December 2014 - February 2015
  Response to survey

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Providence Hospital, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No